CLINICAL TRIAL: NCT01730235
Title: My MediHealth: A Paradigm for Children-centered Medication Management
Acronym: mymedihealth
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kevin Johnson, Professor and Chair, Biomedical Informatics, Vanderbilt University
Other Study IDs: R18HS018168 (AHRQ)
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Group: Group receiving access to MyMediHealth web site.
- Control Group: Children completing baseline and week two measures, but without any additional intervention.
  Interventions: Other: MyMediHealth access

INTERVENTIONS:
Other: MyMediHealth access — Patients who will be given access to a web-based medication scheduling and SMS-based reminder system.
  Groups: Control Group

SUMMARY:
The last mile of the medication use system requires tools to help patients comply with medication administration rules and monitor for side effects. Personal health records (PHR) and emerging user-adopted communication tools promise to change the landscape of medication management. The overarching goal of the MyMediHealth project is to investigate ways in which PHRs and supported applications can improve the safety and quality of medication delivery. Preliminary work in this area by a team of parents, patients and school/clinic health providers created a vision for MyMediHealth, a next-generation medication management system. MyMediHealth was envisioned to allow home-based, school-based, and other caregivers to ensure safe and effective medication delivery. This vision featured just-in-time medication reminders to children with special health care needs, two-way communication to log when doses have been administered or when side effects have occurred, and mechanisms to warn caregivers about side effects and drug interactions. However, much of this work was done using prototypes, storyboards, and vision videos. Recognizing that this vision cannot be carried out without significant changes in processes and policies, the purpose of this proposed study is to evaluate the impact of medication management tools such as MyMediHealth on medication adherence for children with chronic illnesses. Specifically, the investigators hypothesize that compared with usual practice, children using mymedihealth will have improved medication adherence and will report improved (decreased) asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Access to the internet Caregiver agrees to let child use the Internet for the project Internet service working properly Legal guardian approves of study Child with her or his own cell phone

Exclusion Criteria:

* non English or spanish speaking family

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescents between the ages of 12 and 17 with a diagnosis of asthma and on at least one daily medication.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline asthma self efficacy after 3 weeks | participants will be followed for an average of 4 weeks, with this measure collect at the beginning of the period and after 3 weeks of reminders.
  Will assess self-efficacy using the survey by Bursch and colleagues (1997)

SECONDARY OUTCOMES:
Change in medication adherence after 3 weeks | Participants will be followed for 4 weeks, with measurements at baseline and the end of 3 weeks
  At the end of the 2-week data collection period (following the 1-week test period), all participants (Control and Intervention) and their parents will be asked to complete a brief online survey, including the Asthma Control Test (ACT) and the weekly adherence survey(SDSCA). All responses collected from participants and their parents in the Time 2 Survey will be compared to those collected from the Baseline Survey, where applicable. Medication adherence will be measured by responses to ACT and SDSCA survey items for all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Vandebilt Monroe Carell Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Johnson KB, Patterson BL, Ho YX, Chen Q, Nian H, Davison CL, Slagle J, Mulvaney SA. The feasibility of text reminders to improve medication adherence in adolescents with asthma. J Am Med Inform Assoc. 2016 May;23(3):449-55. doi: 10.1093/jamia/ocv158. Epub 2015 Dec 11. PMID 26661717